CLINICAL TRIAL: NCT04321837
Title: Coral Calcium's Effect on Bone Density in Postmenopausal Women With and Without Ibandronate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of California, Irvine (Other); Osteoporosis Center of Armenia (Unknown)
Responsible Party: Principal Investigator, John P. Bilezikian, Dorothy L. and Daniel H. Silberberg Professor of Medicine and Professor of Pharmacology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAS2051; HS# 2018-4772 (Other: University of California, Irvine)
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Calcium; Coral calcium; Ibandronate
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Coral calcium complex and ibandronate (Active Comparator)
  Interventions: Dietary Supplement: Coral Complex 3; Drug: Ibandronate
- Ibandronate and vitamin D (Active Comparator)
  Interventions: Drug: Ibandronate; Dietary Supplement: Vitamin D3
- Coral calcium complex (Active Comparator)
  Interventions: Dietary Supplement: Coral Complex 3

INTERVENTIONS:
Dietary Supplement: Coral Complex 3 — Coral-derived calcium supplement fortified with vitamin D3
  Arms: Coral calcium complex; Coral calcium complex and ibandronate
Drug: Ibandronate — Bisphosphonate
  Arms: Coral calcium complex and ibandronate; Ibandronate and vitamin D
Dietary Supplement: Vitamin D3 — Oral vitamin D3
  Arms: Ibandronate and vitamin D

SUMMARY:
This study will investigate the effect of coral calcium complex supplementation on BMD of osteoporotic individuals either when used alone or in combination with ibandronate. Ibandronate alone will also be tested in comparison to coral calcium supplementation alone or in combination.

DETAILED DESCRIPTION:
Osteoporosis and resulting fragility fractures are major causes of morbidity and mortality in older individuals. Current estimates indicate that as many as 50% of American women and 20% of men over the age of 50 will be at risk for osteoporotic fractures during their lifetimes, and that these fractures are associated both with higher risk for further fractures and with higher mortality rates. Osteoporosis and subsequent fragility fractures can be prevented if diagnosed and treated appropriately. The first step of treatment guidelines for individuals with reduced bone mineral density (BMD), as identified with dual energy x-ray absorptiometry (DXA) scan, is the implementation of lifestyle measures to reduce bone loss. These include the supplementation of dietary calcium and vitamin D to maintain appropriate calcium intake and reduce resorption of mineralized calcium from bone. Pharmacological treatment can be used for the treatment of osteoporosis in individuals who have reduced BMD (less than -2.5 T-score) and for those who have sustained a fragility fracture. The bisphosphonates are first line agents for the treatment of osteoporosis. Coral-derived calcium is a novel formulation of calcium supplement, which has not yet been rigorously investigated as an efficacious nutrient for the skeleton. Ibandronate is a commonly available bisphosphonate prescribed for the treatment of osteoporosis. Vitamin D is a nutrient required to absorb vitamin D from the diet.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women, 50-75 years of age (inclusive). Menopause is defined as no menstrual period for 1 year.
2. BMD T-score of lumbar spine (L1-L4), femoral neck, total hip, or non-dominant forearm < -2.5 as determined by DXA.

Exclusion Criteria:

1. T-score of lumbar spine, femoral neck, total hip, or non-dominant forearm < -3.5.
2. Use of any supplemental calcium preparations in the past 1 year.
3. Use of ibandronate in the past 3 years.
4. Current use of

   1. prednisone or other corticosteroid,
   2. antiseizure medications,
   3. thiazide diuretics, or
   4. estrogen preparation except vaginal cream.
5. Electrolyte abnormalities, as defined by abnormal blood levels of sodium (Na), chlorine (Cl), potassium (K), phosphate (Phos), calcium (Ca), or magnesium (Mg) values on initial screen.
6. Chronic disease, including

   1. liver disease (as defined by elevated blood levels of aspartate aminotransferase, alanine aminotransferase, and/or alkaline phosphatase or reduced albumin or total protein on initial screen),
   2. stage III renal disease or worse (as defined by epidermal growth factor receptor (eGFR) < 60 cc/min),
   3. abnormal thyroid function tests,
   4. current parathyroid disease (as defined by hypercalcemia and elevated levels of parathyroid hormone (PTH) - if history of hyperparathyroidism, surgical cure has to be documented more than 5 years ago),
   5. diabetes mellitus,
   6. any other known metabolic bone disease besides osteoporosis, and/or
   7. any inflammatory, anatomic, or malabsorptive GI tract disease.
7. Osteoporotic fracture in the past 6 months, defined as a low-energy fracture such as a fracture after falling from a standing height.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Mean change in bone mineral density (BMD) (lumbar spine) | 48 weeks
  Participant bone mineral density of lumbar spine.
Mean change in BMD (femoral neck) | 48 weeks
  Participant bone mineral density of femoral neck.
Mean change in BMD (total hip) | 48 weeks
  Participant bone mineral density of total hip.
Mean change in BMD (forearm) | 48 weeks
  Participant bone mineral density of forearm.

CONTACTS AND LOCATIONS:
Overall Officials: John P Bilezikian, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Osteoporosis Center of Armenia, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: No